CLINICAL TRIAL: NCT04881773
Title: Oral Low Doses Tolerance INduction Study for Peanuts
Acronym: OLDTINYpeanut
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0254
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Peanut Allergy
Keywords: Food allergy; peanuts; Oral Immunotherapy; efficacy; safety; Peanut IgE mediated allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several protocols have been proposed in scientifis literature, for oral tolerance induction (OIT) protocols for peanuts. A meta-analysis showed that the data in the literature are rather in favor of the exclusion of peanuts, and that OIT doesn't allow to expect significant levels of peanut protein consumed by the patient, and is associated with an increased risk of anaphylaxis and epinephrine use. Also, in most published protocols, patients with a history of anaphylactic shock, severe asthma, or multiple history of anaphylaxis are excluded.

To date, no protocol has been validated for this type of treatment, and each center follows locally validated schemes. In our unit, the investigators use an OIT protocol that starts at low doses (first dose at 2.68 mg peanut protein) and doses increase is scheduled every 4 to 12 weeks (instead of every 2 weeks). The investigators do not exclude patients with asthma or those with a history of peanut anaphylaxis (grade 2 or 3). The investigators have noted that our protocol is associated with a good safety profile and good efficacy, probably due to the fact that the investigators start at low doses and increase the dose with a prolonged delay, compared to previously published protocols. For this reason, the investigators decided to evaluate the results the investigators obtained in our patients and to better analyze the efficacy and safety profile of our protocol.

ELIGIBILITY:
Inclusion criteria:

* Patients evaluated at the Montpellier University Hospital, Allergy Unit ;
* Patients aged 5 years or older;
* Patients with a history of immediate reaction after consuming peanuts
* AND a positive peanut prick test;
* AND peanut positive specific serum IgE (ImmunoCAP®);
* AND a positive oral peanut challenge test OR a clinical history of anaphylaxis AND peanut-specific IgE> 100 kUA / L (ImmunoCAP®);
* Patients who started peanut OIT between September 2018 and January 2021.

Exclusion criteria:

* Patients in exclusion period determined by a previous study;
* Patients under legal protection, under guardianship or under curatorship;
* Possible poor therapeutic compliance to the OIT protocol;
* Active malignant neoplasia or autoimmune disease;
* Active eosinophilic esophagitis or other gastrointestinal eosinophilic disorders;
* Severe active eczema;
* Pregnancy ;
* Cardiovascular disease and use of beta blockers and / or ACE inhibitors;
* Chronic urticaria;
* Mastocytosis.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older that 5 years of age, with a diagnosis of IgE mediated peanuts allergy, undergoing a oral immunotherapy protocol for peanuts, at the University Hospital of Montpellier (France)
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who reach a tolerated dose | 24 months
  Percentage of patients who reach a tolerated dose of 2000 mg of PP during the ITO and percentage of patients who reach a cumulative tolerated dose of 4400 mg of PP during the oral challenge, carried out at least 6 month after the end of the ITO.

SECONDARY OUTCOMES:
Percentage of patients experiencing side effects during OIT | 24 months
  Percentage of patients experiencing side effects during OIT (classified on the basis of their severity); percentage of patients in whom the tolerated dose of PP could be doubled and tripled, compared to the eliciting dose, assessed during an oral food challenge before the beginning of the OIT; percentage of patients who achieve a tolerated dose of 300 mg of PP and 1000 mg of PP during OIT. By doing a subgroup analysis, we will evaluate the same results in patients with a clinical history of grade 2 or grade three anaphylaxis to peanuts.

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC